CLINICAL TRIAL: NCT01692249
Title: Spa Therapy in the Treatment of Chronic Shoulder Pain Due to Rotator Cuff Tendinopathy: ROTATHERM, a Large Randomized Multicentre Trial
Brief Title: Efficacy and Safety of Spa Treatment in Chronic Shoulder Pain Due to Rotator Cuff Tendinopathy
Acronym: ROTATHERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFRETH 2
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Self Efficacy
Keywords: chronic shoulder pain; rotator cuff tendinopathy; sap therapy; balneotherapy
MeSH Terms: interventions — Balneology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate spa therapy (Experimental): group (A) received immediate spa treatment, with 18 days of therapy over 3 weeks; The standardized shoulder therapy program was designed by experienced spa therapy physicians. Spa mineral water and treatments are approved and controlled by the French authorities. Spa treatment included: bubble buses at 36°C for 15 minutes, applications of mineral matured mud at 45°C to the shoulder for 20 minutes, mineral hydrojet sessions at 39°C for 7 minutes and general mobilization in a collective mineral water pool at 35°C for 20 minutes supervised by a registered physiotherapist.
  Interventions: Other: immediate spa therapy
- control group (No Intervention): in group (B), spa therapy was delayed for 6 months (control group).

INTERVENTIONS:
Other: immediate spa therapy — , with 18 days of therapy over 3 weeks; The standardized shoulder therapy program was designed by experienced spa therapy physicians. Spa mineral water and treatments are approved and controlled by the French authorities. Spa treatment included: bubble buses at 36°C for 15 minutes, applications of mineral matured mud at 45°C to the shoulder for 20 minutes, mineral hydrojet sessions at 39°C for 7 minutes and general mobilization in a collective mineral water pool at 35°C for 20 minutes supervised by a registered physiotherapist.
  Other Names: spa treatment; balneotherapy; physical treatment
  Arms: immediate spa therapy

SUMMARY:
To determine whether spa therapy has a beneficial effect on pain and disability in the management of shoulder pain due to chronic rotator cuff lesions, this multicentre randomized prospective clinical trial includes patients with shoulder pain due to chronic degenerative rotator cuff tendinopathy who attend French spa resorts as outpatients. Subjects are randomized into two groups: immediate spa therapy (18 days of standardized treatment) and control (spa therapy delayed for 6 months). All patients continue usual treatments during the 6-month follow-up period. The main endpoint is the mean change in the DASH score at 6 months. Secondary endpoints are the mean change in SF-36 components, treatments used, and tolerance. The effect size of spa therapy is calculated and the proportion of patients reaching minimal clinically important improvement (MCII) is compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic shoulder pain (symptom duration of more than 6 months) due to primary or secondary tendinopathy of the rotator cuff.

In cases of rotator cuff tendinopathy related to traumatic events, the trauma was required to have happened at least 6 months previously. Corticosteroid treatment for concomitant disease could be continued at a stable dose. Shoulder x-rays within the previous 18 months were required in all cases.

Exclusion Criteria:

* shoulder pain related to neurological or vascular disorders or neoplasms; referred pain from internal organs; systemic rheumatic conditions; inability to complete questionnaires because of cognitive impairment, or language difficulty; contraindication (immune deficiency, evolving cardiovascular conditions, cancer, infection, non-equilibrated diabetes mellitus) or intolerance to any aspect of spa treatment; spa treatment within the previous 6 months; steroid injection within the previous 3 months; physiotherapy in the previous month; changes in non-steroidal anti-inflammatory drug (NSAID) administration within the previous 5 days or in other analgesic drug use within the previous 12 hours.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
changes in the Disability of arm, shoulder and hand score (DASH) between baseline and 6 months | self-reported patient outcomes
  The domains explored by the Quick DASH are: (1) physical arm, shoulder or hand activity problems (6 items); (2) severity of pain and tingling (2 items); (3) social activities, work, and sleep (3 items). Each item has five response options, ranging from 1, ''no difficulty or no symptom,'' to 5, ''unable to perform activity or very severe symptom.'' If at least 10 of the 11 items are completed, a score ranging from 0 (no disability) to 100 (most severe disability) can be calculated [(sum of n responses/n) - 1] x 25.the effect size and the percentage of patients reaching Minimal Clinical Important Improvement was determined

SECONDARY OUTCOMES:
changes in the Short-form 36 questionnaire (SF-36) between baseline and 6 months | self-reported patient outcomes
  The SF-36 is the most widely used generic instrument for assessing physical, mental, and psychosocial health based on eight scales and two component summary scales (Physical and Mental Component Summary) containing a total of 36 items
adverse and severe adverse events | recording of SAE and AE
  all SAE and AE were recorded during the spa therapy and the 6-month follow-up
changes in treatment consumption between baseline and 6 months | All treatments were self-recorded by patients.
  analgesics, analgesics plus NSAIDs, rehabilitation and topical medications were recorded during the 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Gay, MD,PhD, Study Director — Association Francaise pour la Recherche Thermale
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Result] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131